CLINICAL TRIAL: NCT05662241
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Obexelimab in Patients With IgG4-Related Disease (INDIGO)
Brief Title: A Phase 3 Study of Obexelimab in Patients With IgG4-Related Disease
Acronym: INDIGO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB012-03-001
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: IgG4 Related Disease
Keywords: IgG4; IgG4-RD
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZB012 (Experimental): Obexelimab administered as an SC injection.
  Interventions: Drug: Obexelimab
- Placebo (Placebo Comparator): Placebo administered as an SC injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Obexelimab — Obexelimab is a monoclonal antibody that co-engages CD19 and FcγRIIb to inhibit B cell activity
  Arms: ZB012
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to examine the efficacy and safety of obexelimab for the prevention of flare of IgG4-related disease (IgG4-RD)

DETAILED DESCRIPTION:
This study consists of a 1-year randomized control period (RCP), followed by an additional 3-year open label extension (OLE) period.

To enter the Screening Period (Day -28 to Day -1), patients must have active IgG4-RD signs/symptoms (i.e., flare) that require steroid therapy. On Day 1, patients will be randomized in a ratio of 1:1 to receive either obexelimab or placebo administered as subcutaneous (SC) injections. All patients will begin a steroid taper on Day 1 to discontinuation by Week 8.

Patients will be monitored for flares during scheduled in clinic visits and any unscheduled visits. The primary endpoint is time to first IgG4-RD flare that requires initiation of rescue therapy in the opinion of the investigator and the Adjudication Committee (AC).

Following the 52-week RCP, patients will have the opportunity to continue in an OLE period where all patients will receive obexelimab. During the OLE, a subset of patients may be eligible to participate in a sub-study evaluating the immune response to vaccination while receiving obexelimab treatment. Patients who do not wish to enroll into the OLE period will return for an in-clinic safety follow-up visit 8 weeks after the Week 52 visit (i.e., Week 60).

Including screening and follow-up, the maximum duration of participation in this study for an individual patient is 224 weeks (i.e., 28-day screening, 52-week RCP, 156-week OLE, and a 12-week follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥ 18 years of age
2. Clinical diagnosis of IgG4-RD
3. Patients must meet the 2019 ACR/EULAR Classification Criteria for IgG4-RD
4. Patients must have active IgG4-RD signs/symptoms (i.e., flare) that require the initiation of GC therapy or the increase in background long-term GC therapy
5. Other inclusion criteria apply

Exclusion Criteria:

1. Has disease in only 1 organ system whose primary manifestation is fibrosis
2. Has received prednisone equivalent given orally at a dose greater than 60 mg/day within the 4 weeks prior to screening or during screening
3. Has received a non-biologic, disease-modifying anti-rheumatological drug or immunosuppressive agent other than GCs within the 2 weeks prior to screening
4. Has received an investigational treatment or direct medical intervention on another clinical study within 12 weeks or < 5 half-lives of the investigational treatment, whichever is shorter, prior to screening
5. Has received live vaccine or live therapeutic infectious agent within the 2 weeks prior to screening
6. Active tuberculosis or high risk for tuberculosis; hepatitis C infection in absence of curative treatment; evidence of hepatitis B infection
7. Use of B cell depleting or targeting agents within 6 months of randomization
8. Other exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | Randomization to Week 52
  Time to first IgG4-RD flare, defined as the reappearance of previous signs/symptoms or appearance of new signs/symptoms of IgG4-RD that requires initiation of rescue therapy in the opinion of the investigator and the Adjudication Committee (AC), from randomization to Week 52.

OTHER OUTCOMES:
Vaccine antibody titers | During the 3 year OLE period
  Vaccine antibody titers at multiple timepoints post-vaccination

CONTACTS AND LOCATIONS:
Locations (65):
- United States (5):
  - Stanford Medicine, Stanford, California
  - GI PROS Research - Dedicated Research Facility, Naples, Florida
  - Emory Univeristy, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Canada (3):
  - Artus Health Centre, Vancouver, British Columbia
  - Center for Clinical Research (Nova Scotia Health), Halifax, Nova Scotia
  - Centre Hospitalier Universitaire de Sherbrooke CHUS, Sherbrooke, Quebec
- China (9):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhai, Hubei
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
- France (4):
  - Haut-Lévèque Hospital Usn Building South Hospital Group, Pessac, Bordeaux
  - Hôpitaux Universitaires de Marseille Timone, Saint-Pierre, Marseille
  - Hôpital Beaujon, Paris
  - Hôpital de la Pitié Salpétrière, Paris
- Germany (2):
  - LMU Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Ulm, Ulm
- Italy (5):
  - Ospedale San Giovanni Bosco, Turin, Piedmont
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Meyer Istituto di Ricovero e Cura a Carattere Scientifico, Florence
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - University of Verona, Verona
- Japan (20):
  - Hospital of University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Kanazawa Medical University Hospital, Kokura, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Hiragi, Kagawa-ken
  - Shinshu University Hospital, Matsumoto, Nagano
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - The Institute of Medical Science, The University of Tokyo Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - Kansai Medical University Hospital, Hirakata
  - Hiroshima University Hospital, Hiroshima
  - St. Marianna University Hospital, Kawasaki
  - Tokyo Medical Center Hospital, Meguro City
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki University Hospital, Nagasaki
  - Kita-Harima Medical Center, Ono
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka
  - Sapporo Medical University Hospital, Sapporo
  - Fujita Health University Hospital, Shinjuku-Ku
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Centro de Alta Especialidad En Reumatologia E Investigacion Del Potosi SC, San Luis Potosí City
- Poland (2):
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw, Masovian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
- South Korea (2):
  - Seoul National University Hospital, Seoul, Seoul
  - Ajou University Hospital, Suwon
- Spain (4):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Medicine, Altındağ, Ankara
  - Marmara University Pendik Training and Research Hospital, Pendik, Istanbul
- John Radcliffe Hospital, Oxford, United Kingdom